CLINICAL TRIAL: NCT01116570
Title: Exercise and Myopathies. Physical Training Introduction in Lifestyle of Facioscapulohumeral Dystrophy Patients: Functional, Tissue and Quality of Life Benefits.
Brief Title: Physical Training Introduction in Lifestyle of Facioscapulohumeral Dystrophy Patients
Acronym: FSHD1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Association Française contre les Myopathies (AFM), Paris (Other); Örebro University, Sweden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1001035; 2010-A00288-31 (Other: AFSSAPS); 2009.1087-14263 (Other Grant/Funding Number: AFM)
Record Dates: First submitted 2010-04-28; First posted 2010-05-05 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Muscular Dystrophy, Facioscapulohumeral
Keywords: Muscular Dystrophy; Facioscapulohumeral; Physical training; Exercise
MeSH Terms: conditions — Muscular Dystrophy, Facioscapulohumeral; Muscular Dystrophies; Motor Activity | interventions — Physical Conditioning, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical training (Experimental): The training will consist in 3 sessions of 35 min of training per week at home on an ergocycle. As a result, lower limb muscles will be mainly solicited. These muscles are heterogeneous in terms of deficiency, but this latter is compatible with cycling. The training will be divided in (i) 2 sessions of 30 min aerobic exercises at a constant but moderate (60% of maximal aerobic power, MAP) intensity followed with 5 sets of 10 revolutions at near-maximal intensity and (ii) an interval-training session. This latter session will consist in 5 min warm-up at 40% MAP followed by 5 times 1 min at 80% MAP (recovery = 4 min at 40% MAP) followed by 5 min of active recovery. Over a 2 to 4 weeks initial period, the program will be conducted in the laboratory or at home under the supervision of a coach. Then a systematic supervision of the sessions by the coach will be performed by phone, by using the heart rate recordings and values of Analogic Visual Scale for pain and fatigue.
  Interventions: Other: Physical training
- control (Other): None intervention
  Interventions: Other: Control

INTERVENTIONS:
Other: Physical training — Physical training during 24 weeks
  Arms: Physical training
Other: Control — No intervention
  Arms: control

SUMMARY:
It is now accepted that physical activity is not deleterious in myopathies, including muscular dystrophies. In patients suffering from facioscapulohumeral dystrophy (FSHD), aerobic training has been reported to be associated to physiological and functional positive effects without alteration in quality of life. The review papers from Van der Kooi et al. (2005), Cup et al. (2007) and Féasson et al. (2010) suggest that the combination of endurance and strength training is even more relevant. Only a few controlled and randomized studies have been conducted on this topic. The impact of such training programs on the skeletal muscle regenerative capacities has not been yet addressed. Moreover, due to the fact that training programs are mainly performed on short-term supervised periods, there is a lack of knowledge regarding long-term effects, patient's autonomy and whether or not regular exercise practice can be maintained in patient's daily life. Also, only a few experiments have reported an integrative view of the potential benefits of such programs on functional, biological and quality of life.

DETAILED DESCRIPTION:
Our research project aims at establishing a program of physical training that will fulfill the two following conditions: (i) being compatible with the daily professional, social and family activity of the patients so it can be integrated in their life habits and (ii) being intensive enough to induce functional benefits. This experimental work will be based on multi-factorial evaluations, i.e. biological, physiological, functional, and quality of life questionnaires. This work will be based on a collaboration between the Universities of Saint Etienne (L. Féasson), Grenoble (B Wuyam) and Örebro (F Kadi) within the Rhône-Alpes Reference Centre for Rare Neuromuscular Diseases (JC Antoine).

It is accepted that exercise therapy can be recommended for patients with myopathies but long-term training load still has to be determined for each pathology. In the specific context of facioscapulohumeral dystrophy, we aim at associating the scientific evaluation of physical activity benefits and a therapeutic education of patients in order to contribute to recommendations for physicians and physiotherapists. The purpose of this study is to combine an integrated approach with a better understanding of biological process implicated in this physiological treatment strategy.

ELIGIBILITY:
Inclusion Criteria:

* facioscapulohumeral dystrophy
* Being capable of supporting an exercise on ergocycle
* Social Security regimen affiliated
* Consent form signed

Exclusion Criteria:

* Severe cardiac or respiratory insufficiency
* Cardiac pacemaker
* Morbid obesity (BMI upper to 35)
* Anti platelet therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-10; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
maximal oxygen uptake (VO2max) | Week 24
  VO2max is meseasured directly by respiratory gas analysis during maximal exercise test on ergocycle

SECONDARY OUTCOMES:
Questionnaire of quality of life | Day 0, Week 6, Week 12, Week 18 and Week 24
  "short form 36 health survey questionnaire" SF36
Biopsy | Day 0 and Week 24
  biopsy of the vastus lateralis muscle
maximal oxygen uptake (VO2max) | Week 6, Week 12 and Week 18
  VO2max is meseasured directly by respiratory gas analysis during maximal exercise test on ergocycle
Questionnaire of subjective fatigue | Day 0, Week 6, Week 12, Week 18 and Week 24
  Fatigue severity scale (FSS)
nuclear magnetic resonance imaging | Inclusion
  In Paris centre, a total body NMR imaging will be done with standard T2- and T1-weighted images.

CONTACTS AND LOCATIONS:
Overall Officials: Leonard FEASSON, MD-PhD, Principal Investigator — CHU de Saint-Etienne; Fawzi KADI, MD-PhD, Study Chair — Orebro University, Sweden
Locations (2):
- France (2):
  - CHU de Grenoble, Grenoble
  - CHU de Saint-Etienne, Saint-Etienne